CLINICAL TRIAL: NCT04641377
Title: A Multicomponent Exercise Intervention Using Telehealth to Improve Psychological and Physical Outcomes in Breast Cancer Patients Undergoing Primary Treatment: A Randomized Controlled Trial
Brief Title: Adaptations to Breast Cancer and Exercise Using Telehealth (ABRACE: Telehealth)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Stephanie Santana Pinto, Principal investigator, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CAAE: 39277420.8.0000.5313
Record Dates: First submitted 2020-11-12; First posted 2020-11-23 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent exercise intervention plus health education (Experimental): The multicomponent training will be performed twice a week, on pre-established and non-consecutive days. The sessions will be held by video call (approximately 60 min) in small groups (maximum three participants) and will be taught by students of the Physical Education course, previously trained to carry out the intervention. The order of the multicomponent training will be: joint mobilization, aerobic stimulus, balance exercise, strength exercises and stretching of the main muscles used during the training session. Health education will also be carried out on one of the two days. The conversation on the topic of the week will take place during stretching.
  Interventions: Other: Multicomponent exercise intervention plus health education
- Health education (Active Comparator): Once a week, participants in the health education group will be sent a message with a material with various topics related to the management of breast cancer diagnosis and physical activity. In addition, two days after this material is sent, members of ABRACE: Telehealth will have a conversation with the participants of this group, at a google meet of approximately 30 minutes, about the theme sent by message. The themes will be: depression, pain, fatigue, body image, symptoms in the arm and breast, vasomotor symptoms, neuropathy, arthralgia, sexual dysfunction, quality of life, physical activity and eating habits.
  Interventions: Other: Health Education

INTERVENTIONS:
Other: Multicomponent exercise intervention plus health education — The multicomponent training will be performed twice a week, on pre-established and non-consecutive days. The sessions will be held by video call (approximately 60 min) in small groups (maximum three participants) and will be taught by students of the Physical Education course, previously trained to carry out the intervention. The order of the multicomponent training will be: joint mobilization, aerobic stimulus, balance exercise, strength exercises and stretching of the main muscles used during the training session. Health education will also be carried out on one of the two days. The conversation on the topic of the week will take place during stretching.
  Arms: Multicomponent exercise intervention plus health education
Other: Health Education — Once a week, participants in the health education group will be sent a message with a material with various topics related to the management of breast cancer diagnosis and physical activity. In addition, two days after this material is sent, members of ABRACE: Telehealth will have a conversation with the participants of this group, at a google meet of approximately 30 minutes, about the theme sent by message. The themes will be: depression, pain, fatigue, body image, symptoms in the arm and breast, vasomotor symptoms, neuropathy, arthralgia, sexual dysfunction, quality of life, physical activity and eating habits.
  Arms: Health education

SUMMARY:
The aim of the present study is to determine the effects of 12 weeks of multicomponent training associated with a health education program carried out remotely, compared to a health education-only program, on psychological and physical outcomes of women in primary treatment for breast cancer. For that, 36 women will be randomized to a multicomponent training group carried out remotely associated with health education or health education group. The psychological and physical outcomes will be measured pre (week 0) and post-intervention (week 13) in both groups, always by the same investigator blinded in relation to the groups. The multicomponent training group will carry out an exercise program twice a week, and health education will also be carried out on one of the two days. In this group, the conversation on the topic of the week will take place during stretching. The sessions (on pre-established and non-consecutive days) will be held by video call (approximately 60 min) in small groups (maximum three participants) and will be given by students of the Physical Education course, previously trained to perform the intervention. The order of the multicomponent training will be joint mobilization, aerobic stimulus, balance exercise, strength exercises and stretching of the main muscles used during the training session. For the participants of the health education group, also, once a week, a material with several topics related to the management of breast cancer diagnosis and physical activity will be sent by message. In addition, two days after this material is sent, a conversation will be held with the participants of this group, at a google meet of approximately 30 minutes, about the theme sent by message. The themes will be depression, pain, fatigue, body image, symptoms in the arm and breast, vasomotor symptoms, neuropathy, arthralgia, sexual dysfunction, quality of life, physical activity and eating habits. To analyze the outcomes collected, it will be used Generalized Estimating Equations (GEE) and the Bonferroni post-hoc test.

ELIGIBILITY:
Inclusion Criteria:

* Women from the city of Porto Alegre and Pelotas in southern Brazil
* Women diagnosed with breast cancer in stages I-III
* Women undergoing primary treatment (adjuvant or neoadjuvant chemotherapy or only radiotherapy) of breast cancer
* Women can not be practicing periodized and systematic physical exercise programs

Exclusion Criteria:

* Women can not have reached more than 50% of the completion of chemotherapy or only radiotherapy treatment
* Women can not have the following comorbidities:

  * autonomic neuropathy or severe peripheral neuropathy, proliferative diabetic retinopathy, non-proliferative diabetic retinopathy, uncompensated heart failure, unstable angina, peripheral amputations, uncontrolled arterial hypertension, chronic renal failure, severe psychiatric disorders and musculoskeletal impairment that limits physical exercise.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Cancer-related fatigue at 3 months | Baseline and post-intervention (week 13)
  Fatigue will be determined using the behavioural/severity, affective, sensory, cognitive/mood, and total fatigue scores from the Piper Fatigue Scale through an interview. Its version translated into Portuguese is a reliable and valid instrument to measure fatigue in Brazilian cancer patients. This consists of 22 items numerically scaled 0 to 10 that measure the 4 dimensions of subjective fatigue as well as total fatigue.

SECONDARY OUTCOMES:
Change from Baseline Quality of life (QoL) of Cancer Patients at 3 months | Baseline and post-intervention (week 13)
  The impact of cancer and its treatment on QoL will be estimated using the European Organization for Research and Treatment of Cancer (EORTIC) Quality of Life of Cancer Patients (QLQ-C30). The QLQ-C30 is a 30-item questionnaire assessing function and symptoms that impact QoL. It was developed as an integrated measurement system and incorporates 5 functional scales (physical, role, cognitive, emotional, and social: higher scores represent better QoL), 3 symptom scales (fatigue, pain, and nausea and vomiting: higher score corresponds to more frequent and/or more intense symptoms), and 1 global health and QoL scale (higher scores represent better QoL). Several single-item measures assess common cancer symptoms (dyspnea, loss of appetite, sleep disturbance, constipation, and diarrhea: higher score corresponds to more frequent and/or more intense symptoms) and the perceived financial impact of cancer and its treatments.
Change from Baseline Quality of life (QoL) of Breast cancer patients specific supplement at 3 months | Baseline and post-intervention (week 13)
  The European Organization for Research and Treatment of Cancer (EORTIC) breast cancer specific module (QLQ-BR-23), consists of a functional and a symptom scale domains. The scoring algorithm recommended by the EORTC, was used to transform the responses to values on scale 0-100%. For the functional scale, a higher score corresponds to better functioning and HRQOL. For symptom scales, a higher score corresponds to more frequent and/or more intense symptoms. A problematic group is defined as one with a global QoL or functional scale score of 33 or less, and a symptom scale score of 66 or more on the QLQ-BR-23.
Change from Cancer-related cognitive impairment at 3 months | Baseline and post-intervention (week 13)
  The FACT-Cog version 3 comprises 37 items, with four subscales created by the developers: patients' perceived cognitive impairments (CogPCI), perceived cognitive abilities (CogPCA), deficits observed or commented on by others (CogOth), and impact of cognitive changes on quality of life (CogQOL). A global or summary score is obtained by summing all item scores. Respondents indicate the frequency of each occurrence over the 7 days preceding the test on a 5-point Likert-type scale ranging from 0 (never) to 4 (several times per day) in CogPCI and CogOth. In the CogPCA and CogQOL subscales, the responses are rated on a 5-point severity scale ranging from 0 (not at all) to 4 (very much). The individual subscale scores are summed to determine the FACT-Cog total score, ranging from 0 to 132, with higher scores indicating better cognitive functioning.
Change from Depressive symptoms at 3 months | Baseline and post-intervention (week 13)
  The CES-D measures symptoms of depression and is not a diagnostic tool for major depressive disorder. Participants scoring ≥16 (range 0-60) will be considered at risk for prevalent depression. Individuals will be coded as positive for depression if they have a CES-D score of ≥16 and/or had self-report of depression diagnosis at baseline. In addition to the total score, the CES-D includes 4 subscales: depressed affect (range 0-21), positive affect (range 0-12), somatic (range 0-21), and interpersonal (range 0-6).
Change from Anxiety at 3 months | Baseline and post-intervention (week 13)
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. It also is often used in research as an indicator of caregiver distress.Form Y, its most popular version, has 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety. The STAI is appropriate for those who have at least a sixth-grade reading level.
Change from Functional capacity at 3 months | Baseline and post-intervention (week 13)
  The 30-s chair-stand test assesses lower body strength and will be scored by the number of times the participant correctly stands within 30 s. To evaluate upper body strength the arm curl test will be employed. The participant will be instructed to perform as many elbow flexions as possible within a 30-second time limit, always with controlled movements in both the flexion and extension phases. Each complete movement performed correctly will be counted. The tests will be performed with verbal encouragement for all participants, in order to reach their best performance.
Change from Level of leisure-time physical activity at 3 months | Baseline and post-intervention (week 13)
  The Godin-Shephard leisure-time physical activity questionnaire will be used in its validated version and translated into Portuguese in Brazil. Participants should report the number of times per week that they engage in vigorous, moderate and light physical activity for a period of time greater than 15 min. The frequency is multiplied the metabolic equivalent (MET). High scores indicate a higher level of physical activity during leisure.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie S Pinto, PhD, Principal Investigator — Federal University of Pelotas
Locations (2):
- Brazil (2):
  - UFPel, Pelotas, Rio Grande do Sul
  - UFRGS, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Henkin JS, Botton CE, Simon MS, Rocha GG, Silveira CB, Gehrke RS, Freitas GB, Trajano GS, Pinto RS, Pinto SS. Telehealth multicomponent exercise and health education in breast cancer patients undergoing primary treatment: rationale and methodological protocol for a randomized clinical trial (ABRACE: Telehealth). Trials. 2023 Jan 19;24(1):42. doi: 10.1186/s13063-022-07015-z. PMID 36658611